CLINICAL TRIAL: NCT06836908
Title: Chest Compression Synchronized Ventilation (CCSV) - an Exploratory Post Market Clinical Follow-up Study
Brief Title: CCSV - Post Market Clinical Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: WEINMANN Emergency, Medical Technology GmbH & Co. KG (Unknown); Berufsrettung Wien (Unknown)
Responsible Party: Principal Investigator, Sebastian Schnaubelt, MD, Adjunct Professor, Medical University of Vienna
Other Study IDs: CCSV 1
Record Dates: First submitted 2024-05-28; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IPPV: Cardiac arrest patients ventilated with IPPV
- CCSV: Cardiac arrest patients ventilated with CCSV

SUMMARY:
The main goal of this observational study is the evaluation of Chest Compression Synchronized Ventilation (CCSV) regarding oxygenation in terms of PaO2 assessed by routine blood gas analysis, hemodynamic effects, 30-day outcome and safety in comparison to Intermittent Positive Pressure Ventilation (IPPV) as data in humans is sparse especially in direct comparison to other ventilation modes.

Cardiac arrest patients in Vienna, Austria will be preclinically randomized (IPPV and CCSV) and ventilated accordingly during CPR. Differences in oxygenation, decarboxylation, systemic perfusion and cerebral oxygenation, the patient's 30-day outcome as well as ventilator-associated adverse events (e.g., pneumothorax) will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* OHCA
* Correct endotracheal intubation (seen by capnography)
* The patient is being treated by the Vienna Emergency Medical Services within the scope of emergency ventilation.
* MEDUMAT Standard from Weinmann Emergency is used.
* Mechanical ventilation is performed according to the specified indications.

Exclusion Criteria:

* Patients eligible for eCPR (as defined by the standard operating procedure of the Emergency Medical Service Vienna)
* Patients recovering (reaching sustained ROSC) before starting mechanical ventilation or in the first three minutes of it
* Any other mechanical ventilation during the ongoing CPR before study inclusion
* Traumatic cardiac arrest
* Suspected or known pregnancy
* Clinically suspected (tension-)pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult out-of-hospital cardiac arrest patients in Vienna
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Oxygenation | 24 months
  Difference in PaO2 between IPPV and CCSV group

SECONDARY OUTCOMES:
Decarboxylation | 24 months
  Difference in PaCO2 between IPPV and CCSV group
systemic perfusion | 24 months
  differences between IPPV and CCSV in cerebral oxygenation measured by near-infrared spectroscopy (NIRS)
patient outcome | 27 months
  sustained return of spontaneous circulation (ROSC)
ventilator-associated adverse events | 27 months
  Pneumothorax (until hospital admission)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Schnaubelt, MD, PhD, Principal Investigator — Department of Emergency Medicine, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CCSV Whitepaper — https://www.weinmann-emergency.com/fileadmin/data/03_topics/16_ventilation/ccsv/white-paper-ccsv-83701-en.pdf